CLINICAL TRIAL: NCT06999993
Title: Efficacy and Safety of Sodium Hyaluronate Gel Combined With Sodium Bicarbonate Versus Sodium Bicarbonate Alone in Prevention of Failed Back Surgery Syndrome (FBSS)
Brief Title: Efficacy and Safety of Sodium Hyaluronate Gel Combined With Sodium Bicarbonate Versus Sodium Bicarbonate Alone in Prevention of Failed Back Surgery Syndrome
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Misr University for Science and Technology (Other)
Responsible Party: Principal Investigator, Emad Lotfy Mohammed Ahmed, lecturer of Anesthesia & pain, Misr University for Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2022/0098
Record Dates: First submitted 2025-05-22; First posted 2025-05-31 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Postdiscectomy Epidural Fibrosis; Pain
Keywords: Sodium hyaluronate jell; Epidural fibrosis; Sodium bicarbonate; Failed Back Surgery Syndrome (FBSS)
MeSH Terms: conditions — Pain; Failed Back Surgery Syndrome | interventions — orthovisc; Sodium Bicarbonate; Solutions; Injections; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Three parallel groups to compare the effects of different drugs on postdiscectomy epidural fibroses and postoperative pain for 6 months period after surgery
Who Masked: Participant, Outcomes Assessor
Masking Description: the above selected groups are blind regarding the selected intervention drug for each participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Group A (SH): (Sodium Hyaluronate Gel and Sodium Bicarbonate) (n=20) (Experimental): The surgeon will spray the surgical field with 10ml syringe containing 2 ml Sodium Bicarbonate (8.4%), 4 ml Bupivacaine 0.5% and 4ml lidocaine 2%. After that the surgeon will inject Sodium Hyaluronate Gel prefilled syringe (Orthovisc 15mg/ml, 2ml syringe. Anika therapeutics, Inc. 32Wiggins Avenue. Bedford, MA 01730 USA) on the surface of the Dura and the nerve roots before wound closure.
  Interventions: Drug: Sodium hyaluronate jell; Drug: Sodium Bicarbonate
- Group B (SB): (Sodium Bicarbonate) (n=20) (Active Comparator): The surgeon will spray the surgical field with 10 ml syringe containing 2ml Sodium Bicarbonate (8.4%), 4ml Bupivacaine 0.5% and 4ml lidocaine 2% on the surface of the Dura and the nerve roots before wound closure.
  Interventions: Drug: Sodium Bicarbonate
- Group C (control) (n=20) (Placebo Comparator): The surgeon will spray the surgical field with 10ml syringe containing 4ml Bupivacaine 0.5%, 4ml lidocaine 2% and 2ml of saline 0.9% on the surface of the Dura and the nerve roots before wound closure.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Sodium hyaluronate jell — sodium hyaluronate gel was used to decrease or prevent tissue lyres adhesion after surgery
  Other Names: Orthovisc
  Arms: Group A (SH): (Sodium Hyaluronate Gel and Sodium Bicarbonate) (n=20)
Drug: Sodium Bicarbonate — sodium bicarbonate decreases tissue acidosis and so it decreases fibrosis
  Other Names: Sodium bicarbonate 8.4% Solution for Injection
  Arms: Group A (SH): (Sodium Hyaluronate Gel and Sodium Bicarbonate) (n=20); Group B (SB): (Sodium Bicarbonate) (n=20)
Drug: Saline — saline 0.9% is a placebo
  Other Names: saline 0.9%
  Arms: Group C (control) (n=20)

SUMMARY:
This study investigates the efficacy and safety of Sodium Hyaluronate gel combined with Sodium Bicarbonate compared to Sodium Bicarbonate alone in preventing Failed Back Surgery Syndrome (FBSS) and epidural fibrosis after lumbar spine surgery. Will be conducted at Souad Kafafi University Hospital, this randomized controlled trial will involve 60 patients aged 18-70 years scheduled for lumber laminectomy (L4-5 or L5- S1).

60 Patients will be divided into three groups: Group A (n=20) receiving Sodium Hyaluronate and Sodium Bicarbonate , Group B (n=20) receiving Sodium Bicarbonate alone, and Group C (n=20) will be served as the control with saline and local anesthetic. Outcomes will be measured through MRI assessments of epidural fibrosis, pain scores, and satisfaction ratings at 3 and 6 months post-surgery.

DETAILED DESCRIPTION:
Hypothesis:

We hypothesize that Sodium Hyaluronate Jell combined with Sodium Bicarbonate provides a safer and more efficient barrier in preventing Postoperative adhesions in spine surgery than spraying of Sodium Bicarbonate alone on the surface of dura and nerve roots after lumber spine surgery (Laminectomy) for L4-5 and /or L5- S1 disc prolapse.

Ethical Considerations

Before we start the study, we will take approval of the research ethical committee. Informed written consent will be obtained from study participants or their legally authorized representative.

Methodology using

I. Study design

Randomized controlled study

II. Study setting and location

The study will be conducted at the operative theatre of Souad Kafafi University Hospital-Misr University for science and Technology (MUST)

III. Study population:

Patients aged from 18 to 70 years old scheduled for Lumber Spine Surgery (Laminectomy) for L4-5 and/or L5-S1 disc prolapse.

Subjects presenting for Lumber Spine surgery will be randomized in a 1:1:1 ratio to either:

Group A(SH):

Receiving a prefilled syringe with Sodium Hyaluronate Gel after spraying a mixture of Sodium Bicarbonate 8.4%, lidocaine 2% and bupivacaine 0.5% on the surface of dura and nerve roots before closure of the wound.

Group B(SB):

Spraying a mixture of Sodium Bicarbonate 8.4%, lidocaine 2% and bupivacaine 0.5% on the surface of dura and nerve roots before closure of the wound. .

Group C:

Spraying a mixture of lidocaine 2% and bupivacaine 0.5% on the surface of dura and nerve roots before closure of the wound. .

IV. Eligibility Criteria

1. Inclusion criteria

   * Patients scheduled for Lumbar Spine surgery (L4-5 and/or L5-S1 Laminectomy) for disc prolapse.
   * Patients aged >18 years old and below 70 years old.
   * Patients with American Society of Anesthesia (ASA) classification I or II (i.e. ASA classification I: A normal healthy patient, for example: no chronic disease, non-smoking, no or minimal alcohol consumption, BMI<30). (ASA classification II: patients with mild systemic disease, for example: well controlled diabetes/hypertension, smokers, obesity (30 < BMI < 35 )
2. Exclusion criteria

   * Patients aged < 18 years old and above 70 years old.
   * Patients who refuse to participate
   * Patients on Chronic opioid use (addicts, cancer patients receiving palliative treatment,)
   * Patients with ASA classification III or more: patients with life threatening medical conditions, for example: recent myocardial infarction, sepsis, severe cardiac valve dysfunction.
   * Patients with coagulopathy or full anticoagulation.
   * Patients with history of aggressive scar formation.
   * Patients with causes of low back pain other than disc prolapse.
   * Patients with previous lumbar spine surgery.
   * Patients with anemia or acid base disturbances or electrolyte disorders.

V.Study Procedures

1. Randomization Patients will be randomly allocated by a computer-generated table into one of the study groups; the randomization sequence will be concealed in sealed opaque envelopes.
2. Study Protocol

   * All Patients will have a pre-operative assessment visit, which will include; history taking, complete physical examination and review of all the results of the routine investigations (CBC, Coagulation profile, renal functions, liver functions, electrolytes).
   * On Arrival to the preparation room, they will receive the following premedication via intravenous (IV) route: Midazolam 0.03 mg/kg, ondansetron 4 mg & omeprazole 40 mg iv infusion.
   * Upon Arrival to the operating room, the standard Monitoring will be applied which include: Pulse Oximeter, Noninvasive Blood Pressure & Six-lead electrocardiogram (ECG).

The General Anesthesia will be induced using: Propofol 1-2mg/kg, Fentanyl1-2 μg/kg, morphine 0.1mg/kg and Atracurium 0.5 mg/kg. General anesthesia will be maintained using Sevoflurane 1-2 MAC (Mean Alveolar Concentrations) in O2/ Air 50% / 50%, Paracetamol 1gm iv infusion, ketolac 30 mg iv and incremental doses of Atracurium 0.1mg/kg/30 minutes.

At end of the surgery and before wound closure the surgeon will spray the medications on the surface of the dura and nerve roots according to each patient group class.

The patients will be randomly classified into three groups Group A (SH): (Sodium Hyaluronate Gel and Sodium Bicarbonate);

Group B (SB): (Sodium Bicarbonate only);

Group C : control group

VI.Study outcomes

Primary Outcome Measures:

● Grade of epidural fibrosis: as measured by lumbar MRI with contrast at 3 and 6 months after surgery compared with the preoperative lumber MRI.

Scar score ratings will be graded according to the degree of dural scar score in the spinal canal [11]. For each subject, five cross-sectional MR images will be checked, and each cross-sectional image will be divided into four quadrants, so that a total of 20 quadrant cross-sectional MR images per subject will be evaluated.

0= No scar

1. 0-25% of quadrant filled with scar
2. 25-50% of quadrant filled with scar
3. 50-75% of quadrant filled with scar
4. >75% of quadrant filled with scar

Secondary Outcome Measures:

* Postoperative pain score; will be measured by Numerical Rating Scale (NRS) score (0=no pain, 1-3=mild, 4-6=moderate 7-9=severe, 10=most severe) [10]
* Patient and doctor satisfaction with the results of surgery.
* Risk of complications from this technique.

Statistical Analysis

1. Sample size:

   Sample size calculation was based on mean Efficacy and Safety of Sodium Hyaluronate Gel combined with Sodium Bicarbonate in Prevention of Failed Back Surgery Syndrome retrived from previous research ( Ji et al., 2015) [12] . Using G power program version 3.1.9.4 to calculate sample size based on effect size 0.747 ,using 2-tailed test , α error =0.05 and power = 90.0%, the total calculated sample size will be 20 cases at least in each group.
2. statistical analysis: Data will be analyzed using SPSS (statistical package for social sciences) version 22. Qualitative data will be presented as number and percent, Quantitative data will be tested for normality by Kolmogrov-Smironv test then described as mean and standard deviation for normally distributed data and median and range for non-normally distributed. The appropriate statistical test will be applied according to data type with the following suggested tests: Chi-Square for categorical variable, Student t test and Mann Whitney U test for continuous variables.

ELIGIBILITY:
Inclusion Criteria:

This study will include patients scheduled for Lumbar Spine surgery (L4-5 and/or L5-S1 Laminectomy) for disc prolapse, Patients aged >18 years old and below 70 years old and Patients with American Society of Anesthesiologists (ASA) classification I or II.

Exclusion Criteria:

Patients aged < 18 years old and above 70 years old, Patients who refuse to participate, Patients on Chronic opioid use (addicts, cancer patients receiving palliative treatment), Patients with ASA classification III or more, Patients with coagulopathy or full anticoagulation, Patients with history of aggressive scar formation, Patients with causes of low back pain other than disc prolapse, Patients with previous lumbar spine surgery and Patients with anemia or acid base disturbances or electrolyte disorders will be excluded from this study.

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Grade of postoperative epidural fibrosis | one year (20/06/2025 to 31/05/2026)
  ● Grade of epidural fibrosis: as measured by lumbar MRI with contrast at 3 and 6 months after surgery compared with the preoperative lumber MRI.

SECONDARY OUTCOMES:
Chronic postoperative pain | Measured at 3 and 6 months after surgery
  Chronic postoperative pain will be measured by Numerical Rating Scale (NRS) score (0=no pain, 1-3=mild, 4-6=moderate 7-9=severe, 10=most severe)
Risk of complications from this technique | From time of surgery to end of 6 months after surgery
  Risk of epidural infection, nerve root injury, epidural tear or epidural hematoma collection
Patient and doctor satisfaction with surgical results | From time of surgery till 6 months after surgery
  whither satisfied, fair or unsatisfied with the results of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Hany Kamal, prof. of anesthesia, Study Chair — Misr University for Science and Technology (MUST)
Locations (1):
- Souad Kafafi University Hospital (SKUH), faculty of medicine, Misr University for Science and Technology (MUST), Giza, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Demographic Information: Age, sex, race, and other relevant demographic details.
  Baseline Characteristics: Health status, medical history, and any pre-existing conditions prior to the trial.
  Treatment Assignment: Information on the intervention or treatment each participant received.
  Outcome Measures: Data on primary and secondary outcomes as defined in the trial protocol.
  Adverse Events: Reports of any side effects or adverse events experienced by participants during the trial.
  Follow-up Data: Information collected during follow-up periods, including long-term outcomes.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 01/06/2025 to 31/05/2026
Access Criteria: Researchers:
  Who: Academic researchers, industry scientists, and regulatory agencies. What: Full IPD, including demographic data, treatment assignments, and outcome measures.
  How: Through data sharing platforms or repositories after submitting a research proposal and obtaining necessary approvals.
  Regulatory Authorities:
  Who: Agencies like the FDA or EMA. What: Full IPD and supporting documentation for oversight and review. How: Direct access during the review process of clinical trial applications.
  Data Sharing Initiatives:
  Who: Collaborating institutions and consortia. What: Aggregated or anonymized IPD for meta-analyses or systematic reviews. How: Via established partnerships and shared databases.
  Public and Patient Advocacy Groups:
  Who: Organizations seeking to promote transparency. What: Summary data and aggregated results, but not individual-level data. How: Through publicly available reports or dashboards.

REFERENCES:
- [Background] Guyer RD, Patterson M, Ohnmeiss DD. Failed back surgery syndrome: diagnostic evaluation. J Am Acad Orthop Surg. 2006 Sep;14(9):534-43. doi: 10.5435/00124635-200609000-00003. PMID 16959891
- [Background] Epter RS, Helm S 2nd, Hayek SM, Benyamin RM, Smith HS, Abdi S. Systematic review of percutaneous adhesiolysis and management of chronic low back pain in post lumbar surgery syndrome. Pain Physician. 2009 Mar-Apr;12(2):361-78. PMID 19305485